CLINICAL TRIAL: NCT06276010
Title: Use of Nafamostat Mesilate for Anticoagulation in Patients With Extracorporeal Membrane Oxygenation After Cardiac Surgery: Efficacy and Safety
Brief Title: Use of Nafamostat Mesilate for Anticoagulation in Patients With ECMO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xiaotong Hou (Other)
Responsible Party: Sponsor-Investigator, Xiaotong Hou, Clinical professor, Beijing Anzhen Hospital
Organization: Beijing Anzhen Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2023-102
Record Dates: First submitted 2024-02-16; First posted 2024-02-23 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Extracorporeal Membrane Oxygenation Complication
Keywords: anticoagulation; nafamostat mesilate
MeSH Terms: interventions — nafamostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nafamostat mesilate group (Experimental): The initial dosing of the nafamostat mesilate group is 0.5mg/kg/h. We maintain ACT at 180~220s by adjusting the dosage of nafamostat mesilate.
  Interventions: Drug: nafamostat mesilate
- unfractionated heparin group (Other): The initial dosing of the unfractionated heparin group is 8~12U/kg/h. We maintain ACT at 180~220s by adjusting the dosage of unfractionated heparin .
  Interventions: Drug: unfractionated heparin group

INTERVENTIONS:
Drug: nafamostat mesilate — Use nafamostat mesilate as an anticoagulant
  Arms: nafamostat mesilate group
Drug: unfractionated heparin group — Use unfractionated heparin as an anticoagulant
  Arms: unfractionated heparin group

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of nafamostat mesilate compared with unfractionated heparin for anticoagulation in patients with ECMO after cardiac surgery.

DETAILED DESCRIPTION:
Selecting patients who require systemic anticoagulation as the study subjects from patients undergoing extracorporeal membrane oxygenation assistance after cardiac surgery. Randomly divided into the nafamostat mesilate group and unfractionated heparin group. To evaluate the efficacy and safety of nafamostat mesilate by comparing the incidence of bleeding and thrombosis within the target anticoagulant level range between two groups of patients during ECMO

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. VA-ECMO or VV-ECMO was accepted after cardiac surgery.
3. The ECMO treatment team believes that systemic anticoagulation is needed
4. Sign the informed consent form

Exclusion Criteria:

1. The researchers believe that there are other causes of active bleeding that are not suitable to participate in this study.
2. Long-term use of anticoagulants before establishment of ECMO
3. Antiplatelet drugs were used before the establishment of ECMO
4. Severe liver insufficiency
5. Connective tissue disease
6. There is a history of allergy to heparin or nemolastat mesylate.
7. Pregnant
8. Previous diagnosis of heparin-induced thrombocytopenia
9. Expect to die within 48 hours
10. ECPR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of thrombotic complications | Within 7 days after starting anticoagulant therapy
  Thrombotic events include loop thrombosis, oxygenator thrombosis, venous thromboembolism, arterial thromboembolism, and cerebral infarction.

SECONDARY OUTCOMES:
Incidence of severe bleeding complications | Within 7 days after starting anticoagulant therapy
  The definition of bleeding event refers to ELSO Anticoagulation Guideline.
Infusion volume of blood products | Within 7 days after starting anticoagulant therapy
  After randomization, suspended red blood cells, plasma, fibrinogen and platelet volume were infused per person per ECMO day.
ACT qualified rate | Within 7 days after starting anticoagulant therapy
  Number of times ACT detection reached the standard / total number of tests during ECMO
Hospitalization mortality | 28 days
  All-cause mortality
The incidence of oxygenator dysfunction | Within 7 days after starting anticoagulant therapy
  incidence
Heparin-induced thrombocytopenia | Within 7 days after starting anticoagulant therapy
  incidence
Time to reach the target anticoagulant level for the first time | Within 7 days after starting anticoagulant therapy

CONTACTS AND LOCATIONS:
Overall Officials: Zhongtao Du, MD, Study Chair — Beijing Anzhen Hospital
Locations (1):
- Beijing Anzhen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No